CLINICAL TRIAL: NCT00539162
Title: Use of the CA 125 Algorithm for the Early Detection of Ovarian Cancer in Low Risk Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Golfers Against Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ID01-022; RP160145 (Other Grant/Funding Number: CPRIT); U01CA200462 (NIH); P50CA083639 (NIH); NCI-2018-02168 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; CA 125 Algorithm; Cancer Detection; Questionnaire; Survey
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CA 125 Analysis (Experimental): Experimental: CA 125, HE4, HE4 antigen autoantibody complexes, and Osteopontin Analysis Participants will have blood (3-4 tablespoons) drawn for CA125 and other tumor markers.
  Depending on CA-125 level and other tumor markers:
  Blood (3-4 tablespoons) drawn for CA-125 testing and other tumor markers in 1 year.
  Blood (3-4 tablespoons) drawn for CA-125 testing and other tumor markers in 3 months, OR
  Blood (3-4 tablespoons) drawn for CA-125 testing and other tumor markers, and a transvaginal ultrasound in 6 weeks +/- 2 weeks.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires completed at baseline and during each follow up visit.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to evaluate a method involving 4 blood tests called CA-125, HE4, HE4 antigen autoantibody complexes, and osteopontin that may be helpful in the early detection of ovarian cancer in women who are at low risk.

DETAILED DESCRIPTION:
Currently, there is no effective screening to detect ovarian cancer at its earliest stage in low risk women. CA-125 is an FDA approved blood test that may show the presence of ovarian cancer. Researchers have found 3 other blood tests (HE4, HE4 antigen-autoantibody complexes, and osteopontin) that detect ovarian cancers that may be missed by CA125 testing. Results of the 4 blood tests are combined into a Risk of Ovarian Cancer-2 (ROCA2) score to decide whether you need to return for additional bloodwork and or an ultrasound.

If you are eligible to take part in this research study:

* You will have blood (about 3-4 tablespoons) drawn for testing CA-125 and other tumor markers that can detect ovarian cancer.
* You will be asked to complete a questionnaire about your medical and family history. It should take about 20-30 minutes to complete.
* You will be asked to complete a questionnaire about your symptoms. It should take about 10-15 minutes to complete.

Depending on your CA-125 level:

* You will have blood (about 3-4 tablespoons) drawn for testing CA-125 and other tumor markers in 1 year.
* You will have blood (about 3-4 tablespoons) drawn for testing CA-125 and other tumor markers in 3 months, OR
* You will have blood (about 3-4 tablespoons) drawn for testing CA-125 and other tumor markers, and you will have a transvaginal ultrasound (to look at your ovaries and fallopian tubes) in 6 weeks +/- 2 weeks.

An ultrasound test uses sound waves to check the position, size, and shape of the ovaries. During a transvaginal ultrasound, a small probe will be placed in your vagina and used to create and measure sound waves.

Based on the results of the transvaginal ultrasound (if you receive one):

* You and the study doctor will discuss options for further treatment or standard cancer management, OR
* You will have blood (about 3-4 tablespoons) drawn for testing CA-125 and other tumor markers in 3 months.

When you return for your next yearly visit:

* You will be asked to complete the questionnaire about your symptoms.
* You will be asked to complete a follow-up visit survey so that any updates to your personal and family medical history can be recorded. It should take about 10 minutes to complete.

Your blood draw results will be sent to you by letter or e-mail so that you will know when to return for a visit.

If you miss a visit, the study staff may try to contact you by telephone, e- mail, or letter. Visit reminders may also be sent to you by letter or e-mail.

If you are unable to return for visits after 3 years, you will be taken off study. You may continue to take part in this study unless you no longer qualify for the study or you no longer would like to take part in this study.

If you develop ovarian or non-ovarian cancer on this study, researchers will no longer collect blood draws, transvaginal ultrasounds, or questionnaires from you. However, the study team will continue to collect updates in your medical record. This includes slides that will be reviewed from cases of ovarian or non-ovarian cancer that are collected as part of your standard of care.

Length of Study:

You will continue to return for visits depending on the CA-125 level from your last visit. If you are unable to return for visits after 3 years, you will be taken off study. You may continue to take part in this study unless you no longer qualify for the study or you no longer would like to take part in this study.

This is an investigational study. Transvaginal ultrasound scans on this study are performed using FDA-approved and commercially available methods.

Up to 8,000 women will take part in this multicenter study. Up to 2,000 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Female, >/= 50 years old or less than 75 years old.
2. Postmenopausal (>/= 12 months amenorrhea).
3. Have at least one ovary.
4. Cancer-free and have not received any chemotherapy or radiation therapy for >/=12 months prior to enrolling on this study.
5. Willingness to return for CA 125 blood tests annually or earlier if indicated.
6. Willingness to return to undergo transvaginal ultrasound if indicated.
7. Women need to provide the name of a gynecologist or qualified healthcare professional willing to provide appropriate follow-up care if indicated

Exclusion Criteria:

1. Female: Less than 50 years old or older than 75 years at the time of enrollment.
2. Psychiatric or psychological or other conditions which prevent a fully informed consent.
3. Prior removal of both ovaries.
4. Active non-ovarian malignancy.
5. Women who have a history of non-ovarian malignancy will be eligible if they have no persistent or recurrent disease and have not received treatment for >12 months. If they are on SERMS (i.e. tamoxifen or aromatase inhibitors) they will not be excluded. Women maybe undergoing or have had treatment <12 months prior to study entry for basal cell carcinoma only.
6. High risk for ovarian cancer due to familial predisposition as defined by the following: a. Known mutation in BRCA1 of BRCA2. b. Two 1st or 2nd degree relatives of same lineage who have: two ovarian cancers; one ovarian cancer & one pre-menopausal breast cancer; two pre-menopausal breast cancers; one pre-menopausal & one post-menopausal breast cancer. (These conditions can also be met using the patient and one 1st or 2nd degree female relative.) c. Ashkenazi Jewish descent with one 1st degree or two 2nd degree relatives with pre-menopausal breast or ovarian cancer or participant has had pre-menopausal breast cancer. d. 1st or 2nd degree male relative with breast cancer diagnosed at any age. (First degree relative defined as children, siblings and parents. Second degree relative defined as half-siblings, aunts, uncles, nieces, nephews, grandparents, and grandchildren.)
7. Hereditary Nonpolyposis Colorectal Cancer (HNPCC)/Lynch Syndrome: known genetic mutation, presumed HNPCC carrier, Amsterdam criteria.

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2001-07-02 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of increase in CA 125 levels and other tumor markers over time | Based on CA-125 level, 3 options will result: 1) re-draw blood (CA-125) in 1 year, 2) re-draw blood (CA-125) in 3 months), or 3) re-draw blood (CA-125) AND TVUS in 6 weeks +/- 2 weeks.
  [Time Frame: Based on CA-125 level and other tumor markers, 3 options will result: 1) re-draw blood (CA-125 and other tumor markers) in 1 year, 2) re-draw blood (CA-125 and other tumor markers) in 3 months, or 3) re-draw blood (CA-125 and other tumor markers) and TVUS in 6 weeks +/- 2 weeks.]

CONTACTS AND LOCATIONS:
Overall Officials: Denise Nebgen, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (11):
- United States (11):
  - Sylvester Comprehensive Cancer Center, Univ of Miami Miller School of Medicine, Miami, Florida
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Carol G. Simon Cancer Center / Atlantic Health, Morristown, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women's and Infant's Hospital, Providence, Rhode Island
  - The University of Texas at Austin, Austin, Texas
  - University of Texas (UT) Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Women's Hospital of Texas, Obstetrics and Gynecology Associates (OGA), Houston, Texas
  - UT Health Science Center San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Han CY, Lu KH, Corrigan G, Perez A, Kohring SD, Celestino J, Bedi D, Bedia E, Bevers T, Boruta D, Carlson M, Holman L, Leeds L, Mathews C, McCann G, Moore RG, Schlumbrecht M, Slomovitz B, Tobias D, Williams-Brown Y, Bevers MW, Liu J, Gornet TG, Handy BC, Lu Z, Bedia JS, Skates SJ, Bast RC Jr. Normal Risk Ovarian Screening Study: 21-Year Update. J Clin Oncol. 2024 Apr 1;42(10):1102-1109. doi: 10.1200/JCO.23.00141. Epub 2024 Jan 9. PMID 38194613
- See also: M D Anderson Cancer Center — http://www.mdanderson.org